CLINICAL TRIAL: NCT06622863
Title: EFFECTIVENESS OF ORAL HYGIENE INSTRUCTIONS GIVEN BY AI-GENERATED VIDEOS VS. TRADITIONAL APPROACH IN PERIODONTAL PATIENTS
Acronym: OHI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Abeer Hakam, Assistant professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MBRU-OHI
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Gingivitis; Periodontitis
MeSH Terms: conditions — Gingivitis; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (C): Standard oral hygiene instructions will be given verbally by the periodontics res (Active Comparator)
  Interventions: Behavioral: Standard oral hygiene instructions will be given verbally by the periodontics resident
- Test group (T): Avatar-based group will receive oral hygiene instructions from a digital avatar of t (Experimental)
  Interventions: Behavioral: Avatar-based group will receive oral hygiene instructions from a digital avatar of their choice

INTERVENTIONS:
Behavioral: Standard oral hygiene instructions will be given verbally by the periodontics resident — Standard oral hygiene instructions will be given verbally by the periodontics resident
  Arms: Control group (C): Standard oral hygiene instructions will be given verbally by the periodontics res
Behavioral: Avatar-based group will receive oral hygiene instructions from a digital avatar of their choice — Avatar-based group will receive oral hygiene instructions from a digital avatar of their choice
  Arms: Test group (T): Avatar-based group will receive oral hygiene instructions from a digital avatar of t

SUMMARY:
Patients attending Dubai Dental Hospital and requiring nonsurgical periodontal therapy will be invited to take part in the study. Potential participants will be screened and selected based on the inclusion and exclusion criteria

The aims of the randomized controlled trial are:

1. To compare the influence of AI-generated instructions versus traditional methods in improving the oral hygiene habits of patients diagnosed with periodontitis
2. To assess the time and cost effectiveness of applying AI-generated oral hygiene instructions in daily practice
3. To evaluate the level of patients' engagement, preference, and satisfaction with technology-based interactions vs. patient-doctor interaction

Research design

* Prospective, in which participants will be recruited and then followed up throughout a specified period of time.
* Randomized, parallel designed, concurrent controlled trial with participants randomly allocated to either control or test groups.

The study will involve two stages, 1) Digital Avatar creation and 2) Clinical component.

The participants will be randomly allocated to two equal sized groups (30 per group) using computer-generated numbers:

Control group (C): Standard oral hygiene instructions will be given verbally by the periodontics resident.

Test group (T): Avatar-based group will receive oral hygiene instructions from a digital avatar of their choice.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 or over.

Diagnosed with gingivitis or generalized periodontitis, Stage I-IV and Grade A-C.

Good compliance and commitment to attend follow-up review appointments.

Willing to provide informed consent.

Exclusion Criteria:

Received periodontal treatment in the last 12 months.

Received systemic anti-inflammatory or antibiotic treatment in the last 3 months.

History of malignancy, radiotherapy, or chemotherapy.

Pregnant or lactating women.

Use of medication known to cause gingival overgrowth.

Participants that require prophylactic antibiotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-06 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Plaque and bleeding score | At baseline and after 3 months

IPD SHARING:
Plan to Share IPD: Undecided